CLINICAL TRIAL: NCT02627755
Title: GlideScope® vs GlideScope® + aScope® for Managing Difficult Airways. Assessment of a New Procedure for Endotracheal Intubation in Patients With Suspected Difficult Airways
Brief Title: GlideScope® vs GlideScope® + aScope® for Managing Difficult Airways.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Manises (Other)
Collaborators: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ROV-GLI-2015-02
Record Dates: First submitted 2015-11-30; First posted 2015-12-11 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Airway Morbidity; Anesthesia Intubation Complication
Keywords: videolaryngoscopy; difficult airway management

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glide group (Active Comparator): Device: Glidescope® use
  Interventions: Device: Glidescope®
- Glide+aScope group (Experimental): Device: combined use of two airway devices Glidescope® + aScope®
  Interventions: Device: aScope®; Device: Glidescope®

INTERVENTIONS:
Device: aScope® — we use the aScope® as a flexible and dirigible guide to facilitate the passage of the endotracheal tube through the vocal cords.
  Arms: Glide+aScope group
Device: Glidescope® — use of Glidescope® in conventional manner to facilitate endotracheal intubation

SUMMARY:
The use in a combined way of two systems of intubation (Glidescope + aScope) would condition an increase in the success rate of endotracheal intubation maneuver compared to conventional isolated Glidescope use in patients with clinical criteria of difficult airway.

DETAILED DESCRIPTION:
Worldwide, up to 600 patients are estimated to die annually as a result of the complications that occur during tracheal intubation The GlideScope® (videolaryngoscope) is used for endotracheal intubation in patients with difficult airway predictors, in this patients overall success intubation rate is 96%. but success intubation rate at first attempt is only 86%.

Despite this positive rates, due to high comorbidity when intubation fails, both failure rates (inverse of success rate) are impermissible. 14% failure at the first attempt intubation as well as 4% overall intubation failure.

in this study the investigators try to show that new procedure associating aScope® (disposable fiberscope) together with GlideScope® increases the success intubation rate of both ( overall and first attempt).

ELIGIBILITY:
Inclusion Criteria:

* Patients programed for general anesthesia with endotracheal intubation required that presents one or both criteria of difficult airway predictors:
* criteria 1: Arne test >10 (Arne J,1998)
* criteria 2: Ratio between neck circumference and thyromental distance > 4. (Kim WH, 2011)

Exclusion Criteria:

* Patients with mouth opening which does not allow the introduction of video laryngoscope.
* Patients with indication of flexible fiberoptic intubation with awake patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-11-21 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-11-21 (Estimated)

PRIMARY OUTCOMES:
first attempt intubation success rate | through study completion, an average of 1 year.
  first attempt intubation success rate

SECONDARY OUTCOMES:
overall intubation success rate | through study completion, an average of 1 year.
  through study completion, an average of 1 year.
intubation time (in seconds) | through study completion, an average of 1 year
  during anesthetic induction time until inflate pneumo tamponade after tracheal intubation
complications related to intubation | 30 days postoperative
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Rovira Soriano, PhD MD, Study Chair — Hospital de Manises; Guido Mazzinari, PhD MD, Principal Investigator — Hospital de Manises
Locations (1):
- Hospital de Manises, Manises, Valencia, Spain

REFERENCES:
- [Background] Griesdale DE, Liu D, McKinney J, Choi PT. Glidescope(R) video-laryngoscopy versus direct laryngoscopy for endotracheal intubation: a systematic review and meta-analysis. Can J Anaesth. 2012 Jan;59(1):41-52. doi: 10.1007/s12630-011-9620-5. Epub 2011 Nov 1. PMID 22042705
- [Background] Aziz MF, Healy D, Kheterpal S, Fu RF, Dillman D, Brambrink AM. Routine clinical practice effectiveness of the Glidescope in difficult airway management: an analysis of 2,004 Glidescope intubations, complications, and failures from two institutions. Anesthesiology. 2011 Jan;114(1):34-41. doi: 10.1097/ALN.0b013e3182023eb7. PMID 21150569
- [Background] Niforopoulou P, Pantazopoulos I, Demestiha T, Koudouna E, Xanthos T. Video-laryngoscopes in the adult airway management: a topical review of the literature. Acta Anaesthesiol Scand. 2010 Oct;54(9):1050-61. doi: 10.1111/j.1399-6576.2010.02285.x. Epub 2010 Jul 28. PMID 20887406
- [Background] Kim WH, Ahn HJ, Lee CJ, Shin BS, Ko JS, Choi SJ, Ryu SA. Neck circumference to thyromental distance ratio: a new predictor of difficult intubation in obese patients. Br J Anaesth. 2011 May;106(5):743-8. doi: 10.1093/bja/aer024. Epub 2011 Feb 24. PMID 21354999
- [Background] Arne J, Descoins P, Fusciardi J, Ingrand P, Ferrier B, Boudigues D, Aries J. Preoperative assessment for difficult intubation in general and ENT surgery: predictive value of a clinical multivariate risk index. Br J Anaesth. 1998 Feb;80(2):140-6. doi: 10.1093/bja/80.2.140. PMID 9602574
- [Derived] Guay J, Williams SR, Robin F, Ruel M. Effect of Intravenous Dexamethasone on the Regression of Isobaric Bupivacaine Spinal Anesthesia: A Randomized Controlled Trial. Anesth Analg. 2019 Jun;128(6):e100-e103. doi: 10.1213/ANE.0000000000003670. PMID 31094803
- [Derived] Mazzinari G, Rovira L, Henao L, Ortega J, Casasempere A, Fernandez Y, Acosta M, Belaouchi M, Esparza-Minana JM. Effect of Dynamic Versus Stylet-Guided Intubation on First-Attempt Success in Difficult Airways Undergoing Glidescope Laryngoscopy: A Randomized Controlled Trial. Anesth Analg. 2019 Jun;128(6):1264-1271. doi: 10.1213/ANE.0000000000004102. PMID 31094798